CLINICAL TRIAL: NCT01889537
Title: Low Dose Ketamine to Enhance VR Analgesia During Painful Burn Care Procedure.
Brief Title: Low Dose Ketamine VR Analgesia During Burn Care Procedure
Acronym: VRK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, David R. Patterson, PhD. ABPP, Professor, National Institute of General Medical Sciences (NIGMS)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 43329-K
Record Dates: First submitted 2013-05-06; First posted 2013-06-28 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Burn
Keywords: Virtual Reality Ketamine
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VR during burn care with Ketamine (Experimental): Comparing Virtual Reality during burn care with Ketamine
  Interventions: Behavioral: Virtual Reality
- VR durin burn care without Ketamine (Experimental): Comparing virtual reality during burn care without Ketamine.
  Interventions: Behavioral: Virtual Reality

INTERVENTIONS:
Behavioral: Virtual Reality — The patient will receive virtual reality during a burn care procedure

SUMMARY:
The purpose of the research is to see whether a low dose of ketamine, a medication used to reduce pain, enhances the effectiveness of a virtual reality video game, which is used as a form of distraction from pain during a painful burn care procedure.

DETAILED DESCRIPTION:
This study is conducted in a hospital setting. It is a randomized controlled trial comparing the use of virtual reality distraction (VRD) and standard pain medications to the use of VRD, standard pain medications and a single low dose of ketamine as a means to reduce pain during a painful procedure in patients in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Compliant and able to complete questionnaires
* No history of psychiatric disorder
* Not demonstrating delirium, psychosis or any form of Organic Brain Disorder
* Able to communicate verbally
* English-speaking
* IV access already in place

Exclusion Criteria:

* Age less than 18 years
* Not capable of indicating pain intensity
* Not capable of filling out study measures
* Evidence of traumatic brain injury
* History of psychiatric disorder
* Demonstrating delirium, psychosis or any form of Organic Brain Disorder and associated memory problems
* Unable to communicate orally
* Receiving prophylaxis for alcohol or drug withdrawal
* Developmental disability
* Any face/head/neck injuries that interfere with the use of Virtual Reality equipment
* Non-English Speaking
* Extreme susceptibility to motion sickness
* Seizure history
* No IV access already in place

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Graphic Rating Scale (GRS) is a questionnaire consists of three subjective pain ratings, one subjective anxiety rating, and one rating of fun using the 0-10. | 1 day (Immediately following burn care )

CONTACTS AND LOCATIONS:
Overall Officials: David R Patterson, Ph.D., Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States